CLINICAL TRIAL: NCT03950908
Title: Single-bite Versus Double-bite Technique for Mapping Biopsies During Endoscopic Surveillance of Hereditary Diffuse Gastric Cancer: a Single Center, Randomized Controlled Trial
Brief Title: Biopsy Technique for Endoscopic Surveillance of Hereditary Diffuse Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Senior Clinician Scientist. Consultant Gastroenterologist., University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FGCS protocol v.10
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Hereditary Diffuse Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single bite (Other): The single bite technique involved removing the forceps with its specimen after each individual biopsy.
  Interventions: Other: Single bite biopsy technique
- Double bite (Other): The double-bite technique involved taking an initial biopsy, repositioning the forceps, and taking another biopsy from the same area with the initial specimen still on the forceps.
  Interventions: Other: Double bite biopsy technique

INTERVENTIONS:
Other: Single bite biopsy technique — During biopsy collection one specimen will be retrieved during a single passage of the biopsy forceps.
  Arms: Single bite
Other: Double bite biopsy technique — During biopsy collection two specimens will be retrieved during a single passage of the biopsy forceps.
  Arms: Double bite

SUMMARY:
Germline mutation in e-cadherin gene (CDH1) is found in approximately 25% to 30% of individuals fulfilling the clinical criteria for hereditary diffuse gastric cancer (HDGC). Prophylactic gastrectomy is the mainstay of the management of cases with pathogenetic CDH1 mutation. However, some individuals refuse gastrectomy and prefer to delay it for medical or psychosocial reasons. For these patients as well as for those in which a pathogenetic mutation is not found, endoscopic surveillance is recommended. The suggested endoscopic protocol involves targeted as well as 30 random biopsies, which is tedious and time-consuming . In order to save time, two specimens can be taken during a single passage of the biopsy forceps ("double-bite" technique). The aim of this study was to determine the adequacy and utility of the "double-bite" technique in patients undergoing surveillance for HDGC as compared to the standard "single-bite technique".

DETAILED DESCRIPTION:
Previous studies have validated endoscopy, as an efficient tool for initial screening and in selected cases surveillance of families fulfilling the clinical criteria for hereditary diffuse gastric cancer (HDGC). The aim is to detect microscopic foci of in situ or intramucosal signet ring cell carcinoma (SRCC), which are characteristic of early HDGC. Currently, the recommended endoscopic protocol involves targeted biopsies of any suspicious lesion as well as a minimum of 30 mapping random biopsies specimens taken from all anatomic areas of the gastric mucosa, also known as Cambridge endoscopy protocol. However this is a time-consuming and tedious process, which significantly prolongs the duration of the procedure and might reduce patient tolerance. In order to save time two specimens can be taken during a single passage of the forceps ("double-bite" technique).

In order to evaluate the adequacy and utility of the "double-bite" technique, patients undergoing surveillance for HDGC, are randomized to the single-bite vs double-bite arm. Endoscopies are performed according to a standardized protocol. Briefly, a white-light high-resolution endoscope with 85 magnification and a maximal resolution of 7.9 mm (GIF-FQ260Z; Olympus, Tokyo, Japan) is used to examine all anatomic segments of the insufflated stomach. Any abnormalities on white-light endoscopy are recorded and assessed further by narrow-band imaging magnification with or without autofluorescence imaging. Targeted biopsy specimens are taken from identified lesions, and 5 random biopsy specimens are taken in each of the siz gastric anatomical areas (prepylorus, antrum, transitional zone, body, fundus, and cardia). The double-bite technique involves taking an initial biopsy, repositioning the forceps, and taking another biopsy from the same area with the initial specimen still on the forceps. The single bite technique involves removing the forceps with its specimen after each individual biopsy. Time is recorded between the first and last random biopsy. Comfort score is reported after the procedure, according to the modified Gloucester scale. The investigators use Boston Single-Use Radial Jaw™ 4 biopsy forceps with a spike. Biopsy specimens are stained with hematoxylin and eosin and periodic acid-Schiff diastase and are assessed for size and presence of SRCC foci by an upper specialist GI pathologist, who have significant experience in SRCC identification. Any lesions are checked by a second pathologist within the Cambridge Pathology team before reporting. Both pathologists are blinded to study arm.

ELIGIBILITY:
Inclusion criteria:

* Patients in the Familial Gastric Cancer Registry held in Cambridge fulfilling clinical criteria for HDGC.
* Patients willing to undergo at least one upper GI endoscopy with random biopsies according to Cambridge biopsy protocol.

Exclusion criteria:

* Patients who decline evaluation with endoscopy either as a screening or surveillance tool
* Patients on clopidogrel, and/or warfarin for high risk condition and unable to withhold temporarily the medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Identification of signet ring cell carcinoma (SRCC) foci. | 1 year
  Evaluating the diagnostic yield of the double-bite technique, by means of identifying SRCC foci, in comparison to the conventional single -bite arm.

SECONDARY OUTCOMES:
Time to perform biopsy protocol. | 1 year
  Differences between the study arms in terms of time required for biopsy collection
Biopsy size | 1 year
  Differences between the study arms in terms of size of the biopsy specimens
Patients comfort | 1 year
  Differences between the study arms in terms of patient comfort score, during the procedure. Comfort score is reported after the procedure, according to the modified Gloucester scale.
  1: No discomfort - resting comfortably throughout; 2: Minimal. One or two episodes of mild discomfort, well tolerated; 3:Mild. More than 2 episodes of discomfort, adequately tolerated; 4: Moderate. Significant discomfort experienced several times during the procedure; 5: Severe. Extreme discomfort, experienced frequently during the procedure
Dose of sedation. | 1 year
  Differences between the study arms in terms of dose required for sedation

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano di Pietro, MD, Principal Investigator — MRC Cancer Unit.University of Cambridge.
Locations (1):
- MRC Cancer Unit, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Post RS, Vogelaar IP, Carneiro F, Guilford P, Huntsman D, Hoogerbrugge N, Caldas C, Schreiber KE, Hardwick RH, Ausems MG, Bardram L, Benusiglio PR, Bisseling TM, Blair V, Bleiker E, Boussioutas A, Cats A, Coit D, DeGregorio L, Figueiredo J, Ford JM, Heijkoop E, Hermens R, Humar B, Kaurah P, Keller G, Lai J, Ligtenberg MJ, O'Donovan M, Oliveira C, Pinheiro H, Ragunath K, Rasenberg E, Richardson S, Roviello F, Schackert H, Seruca R, Taylor A, Ter Huurne A, Tischkowitz M, Joe ST, van Dijck B, van Grieken NC, van Hillegersberg R, van Sandick JW, Vehof R, van Krieken JH, Fitzgerald RC. Hereditary diffuse gastric cancer: updated clinical guidelines with an emphasis on germline CDH1 mutation carriers. J Med Genet. 2015 Jun;52(6):361-74. doi: 10.1136/jmedgenet-2015-103094. Epub 2015 May 15. PMID 25979631
- [Background] Mi EZ, Mi EZ, di Pietro M, O'Donovan M, Hardwick RH, Richardson S, Ziauddeen H, Fletcher PC, Caldas C, Tischkowitz M, Ragunath K, Fitzgerald RC. Comparative study of endoscopic surveillance in hereditary diffuse gastric cancer according to CDH1 mutation status. Gastrointest Endosc. 2018 Feb;87(2):408-418. doi: 10.1016/j.gie.2017.06.028. Epub 2017 Jul 6. PMID 28688938
- [Background] Fewings E, Larionov A, Redman J, Goldgraben MA, Scarth J, Richardson S, Brewer C, Davidson R, Ellis I, Evans DG, Halliday D, Izatt L, Marks P, McConnell V, Verbist L, Mayes R, Clark GR, Hadfield J, Chin SF, Teixeira MR, Giger OT, Hardwick R, di Pietro M, O'Donovan M, Pharoah P, Caldas C, Fitzgerald RC, Tischkowitz M. Germline pathogenic variants in PALB2 and other cancer-predisposing genes in families with hereditary diffuse gastric cancer without CDH1 mutation: a whole-exome sequencing study. Lancet Gastroenterol Hepatol. 2018 Jul;3(7):489-498. doi: 10.1016/S2468-1253(18)30079-7. Epub 2018 Apr 27. PMID 29706558
- [Derived] Pappas A, Tan WK, Waldock W, Richardson S, Tripathi M, Januszewicz W, Roberts G, O'Donovan M, Fitzgerald RC, di Pietro M. Single-bite versus double-bite technique for mapping biopsies during endoscopic surveillance for hereditary diffuse gastric cancer: a single-center, randomized trial. Endoscopy. 2021 Mar;53(3):246-253. doi: 10.1055/a-1201-3125. Epub 2020 Jul 17. PMID 32679601